CLINICAL TRIAL: NCT06973850
Title: The Impact of the Self-efficacy Building Nursing Program on Foot Self-care Confidence and Perceived Risk of Diabetes-related Foot Complications Among Diabetic Elderly Patients: A Randomized Virtual Based Trial
Acronym: foot self-care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Hashem El-Monshed, Department of Psychiatric and Mental Health Nursing, Faculty of Nursing-Mansoura University, Egypt, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Mans01
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Diabetes; Diabetes Mellitus; Foot Care
Keywords: Foot self-care; Self-efficacy; Diabetes-related foot complications; Virtual nursing intervention
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This study utilizes a randomized controlled trial (RCT) design to investigate the effect of a self-efficacy building nursing program on foot self-care confidence and the perceived risk of diabetes-related foot complications among elderly diabetic patients. The intervention is delivered virtually, making the model particularly relevant in the context of limited mobility and accessibility constraints faced by elderly populations.
  Study Design and Setting The study will be conducted at diabetic outpatient clinics located in Damanhour City, El-Behaira Governorate, Egypt. A total of 120 elderly patients diagnosed with type 2 diabetes mellitus will be recruited through purposive sampling and randomly assigned to either the intervention or control group using a computer-generated randomization sequence to ensure allocation concealment. Each group will comprise 60 participants.
  Interventional Study Model This research adopts a parallel assignment model, with participants randomly assigned in
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Control Group Participants in the control group will receive routine diabetes care as provided by the clinic, which may include brief verbal advice about foot care but no structured educational content or follow-up.
- Intervention (Experimental): Intervention Description
  The Self-Efficacy Building Nursing Program is a structured, theory-based educational intervention grounded in Bandura's Self-Efficacy Theory. It aims to enhance participants' confidence in their ability to perform daily foot self-care behaviors and perceive their risk of complications accurately. The content includes:
  Educational modules on diabetes and foot health.
  Training on daily foot inspection, hygiene, nail and skin care, and appropriate footwear.
  Motivational strategies, goal setting, and problem-solving skills.
  Video demonstrations, live discussions, and Q&A sessions with a diabetes nurse educator.
  The program will be delivered over four weekly virtual sessions, each lasting approximately 45-60 minutes, via a user-friendly telehealth platform (e.g., Zoom or WhatsApp Video). Follow-up support and reminders will be provided through weekly text messages and phone check-ins.
  Interventions: Behavioral: The Self-Efficacy Building Nursing Program

INTERVENTIONS:
Behavioral: The Self-Efficacy Building Nursing Program — Intervention Description
  The Self-Efficacy Building Nursing Program is a structured, theory-based educational intervention grounded in Bandura's Self-Efficacy Theory. It aims to enhance participants' confidence in their ability to perform daily foot self-care behaviors and perceive their risk of complications accurately. The content includes:
  Educational modules on diabetes and foot health.
  Training on daily foot inspection, hygiene, nail and skin care, and appropriate footwear.
  Motivational strategies, goal setting, and problem-solving skills.
  Video demonstrations, live discussions, and Q&A sessions with a diabetes nurse educator.
  The program will be delivered over four weekly virtual sessions, each lasting approximately 45-60 minutes, via a user-friendly telehealth platform (e.g., Zoom or WhatsApp Video). Follow-up support and reminders will be provided through weekly text messages and phone check-ins.
  Arms: Intervention

SUMMARY:
Abstract

Background:

Diabetes-related foot complications are a major cause of morbidity among elderly patients with diabetes, often exacerbated by inadequate self-care practices and low self-efficacy. Innovative, accessible interventions are urgently needed to empower patients in preventive foot care.

Objective:

This study aimed to evaluate the impact of a self-efficacy building nursing program, delivered virtually, on foot self-care confidence and perceived risk of foot complications among elderly diabetic patients.

Methods:

A randomized controlled trial will be conducted with 120 elderly diabetic patients recruited from at the diabetic outpatient clinics at Damanhour City of El-Behaira Governorate, Egypt. Participants will be randomly assigned to either an intervention group (60 participants) receiving the virtual self-efficacy building program or a control group ( 60 participants) receiving no interventions.

Outcomes Evaluation:

Outcomes will be measured at baseline (pretest), and immediately post-interventions (Posttest) using validated scales.

Keywords Self-efficacy, Foot self-care, Diabetes-related foot complications, Elderly patients, Virtual nursing intervention, randomized controlled trial

DETAILED DESCRIPTION:
Objectives:

Primary Objective:

• To evaluate the effectiveness of a self-efficacy building nursing program on improving foot self-care confidence among elderly diabetic patients.

Secondary Objectives:

* To assess the impact of the self-efficacy building program on reducing the perceived risk of diabetes-related foot complications among elderly diabetic patients.
* To compare changes in foot self-care confidence and perceived risk between the intervention group and the control group over time (baseline, post-intervention, and 3-month follow-up).
* To determine the feasibility and acceptability of delivering a self-efficacy-based nursing intervention through a virtual platform to elderly diabetic patients.
* To explore the relationship between improvements in foot self-care confidence and reductions in perceived risk of foot complications following the intervention.

Significance:

This research is significant because it addresses the urgent need to prevent diabetes-related foot complications among elderly patients by enhancing their foot self-care confidence through a virtual, self-efficacy building nursing program. By empowering patients to take control of their foot health, the program can reduce serious complications, hospitalizations, and healthcare costs. The virtual delivery model increases accessibility, especially for those with mobility challenges or living in remote areas, and offers a scalable, theory-driven approach that can inform future chronic disease management strategies. Importantly, the study highlights the potential for technology-based nursing interventions to meet the unique needs of vulnerable elderly populations.

Literature Review Diabetes mellitus is a chronic disease associated with numerous complications, including diabetic foot ulcers, infections, and amputations, which disproportionately affect elderly patients (Armstrong et al., 2017). The risk of developing foot complications increases with age, poor glycemic control, and diminished mobility, making elderly populations particularly vulnerable (Lavery et al., 2006). Foot self-care practices, such as daily inspection, proper hygiene, and appropriate footwear use, are essential for preventing diabetic foot complications (International Working Group on the Diabetic Foot [IWGDF], 2019). However, studies have shown that adherence to recommended foot care behaviors is often low among diabetic elderly patients (Al-Khawaldeh et al., 2012).

Self-efficacy, defined by Bandura (1997) as the belief in one's capabilities to execute behaviors necessary to produce specific outcomes, is a critical determinant of health behavior change. In diabetes management, higher self-efficacy has been associated with improved self-care behaviors, including foot care (Sarkar et al., 2006). Enhancing self-efficacy can thus empower patients to consistently engage in preventive behaviors. Several studies have demonstrated that nursing interventions grounded in self-efficacy theory can effectively improve health outcomes in diabetic patients. Programs that incorporate skills training, goal setting, problem-solving support, and positive reinforcement have been particularly successful (Wu et al., 2011). However, research specifically targeting foot self-care confidence in the elderly is limited.

The use of virtual platforms for delivering health interventions has expanded, especially in response to barriers such as reduced mobility and geographical distance. Virtual programs offer flexibility and accessibility, allowing for consistent patient engagement (Bashi et al., 2020). In diabetes management, virtual education and support interventions have shown promising results in improving self-management behaviors (Liang et al., 2021). Despite the growing evidence supporting self-efficacy-based and virtual interventions in diabetes care, few studies have combined these approaches specifically to address foot self-care among elderly patients. Furthermore, limited research has explored the impact of these interventions on patients' perceived risk of foot complications - a factor that may influence motivation for sustained self-care.

Tools of Data Collection

There are four tools wills used for data collection:

Tool I: Socio-demographic and clinical data structured interview schedule It will be developed by the researchers after literature reviewing and included: Demographic characteristics of the elderly patients such as age, sex, social status, level of education, occupation, and income. As well, medical history will be collected.

Tool II: Foot Care Scale for Older Diabetics The Foot Care Scale for Older Diabetics (FCSOD) is a validated tool designed to assess foot self-care behaviors, confidence in performing foot care, and perceived risk of diabetes-related foot complications among elderly diabetic patients. It covers key areas such as daily foot inspection, hygiene, nail and skin care, footwear practices, and professional care seeking. Items are typically rated on a Likert scale, with higher scores indicating better self-care practices and greater confidence. The FCSOD has demonstrated strong reliability and validity, making it a valuable instrument for both clinical assessments and research studies aimed at improving foot health outcomes in older adults. Its user-friendly format also makes it suitable for elderly populations, whether self-administered or conducted via interviews.

Tool III: Foot Care Confidence Scale (FCCS) The Foot Care Confidence Scale (FCCS) is a specialized instrument developed to measure an individual's self-efficacy, or confidence, in performing foot self-care activities to prevent diabetes-related foot complications. It assesses how confident patients feel about tasks such as inspecting their feet, maintaining proper hygiene, choosing appropriate footwear, and seeking professional help when necessary. The scale typically uses a Likert-type format, with higher scores indicating greater confidence in foot self-care abilities. The FCCS has demonstrated good reliability and validity in diabetic populations and is widely used in both clinical and research settings to guide interventions aimed at enhancing self-management and reducing the risk of serious foot problems.

Tool IV: Foot Risk Screening Questionnaire for People with Diabetes The Foot Risk Screening Questionnaire for People with Diabetes is a structured tool designed to identify individuals at increased risk of developing diabetes-related foot complications, such as ulcers and amputations. It typically assesses key risk factors including a history of foot ulcers, peripheral neuropathy symptoms, peripheral arterial disease, foot deformities, and poor glycemic control. The questionnaire gathers patient-reported information and clinical observations, helping healthcare providers quickly stratify patients into different risk categories for appropriate preventive care. It is widely used in clinical practice and research to facilitate early intervention, guide patient education, and prioritize referrals to specialized foot care services, ultimately aiming to reduce the incidence of severe diabetic foot outcomes.

Tool V: Perceived Risk of Amputation Evaluation Form The Perceived Risk of Amputation Evaluation Form is a specialized tool designed to assess how individuals with diabetes perceive their personal risk of experiencing a lower limb amputation due to foot complications. It typically includes items that measure patients' awareness of risk factors, such as poor foot care practices, previous foot ulcers, neuropathy, and poor circulation. Responses are usually recorded on a Likert scale, reflecting levels of concern or perceived vulnerability. This form helps healthcare providers understand patients' risk perceptions, which is important because higher perceived risk can motivate better preventive behaviors. It is often used in research and clinical practice to evaluate the psychological and behavioral aspects influencing diabetic foot care and to tailor educational or intervention programs accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Adults aged 60 years and above.

Diagnosed with type 2 diabetes for at least one year.

Able to use a smartphone or device with internet access.

Willing to participate in a virtual education program.

No current foot ulcers or advanced diabetic foot complications.

Exclusion Criteria:

Cognitive impairment or psychiatric illness affecting comprehension.

Severe visual or hearing impairments preventing participation.

Participation in another educational or foot care intervention study within the past six months.

Exclusion Criteria:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-06-09 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Foot Care Scale for Older Diabetics | through study completion, an average of 1 year
  The Foot Care Scale for Older Diabetics (FCSOD) is a validated tool designed to assess foot self-care behaviors, confidence in performing foot care, and perceived risk of diabetes-related foot complications among elderly diabetic patients. It covers key areas such as daily foot inspection, hygiene, nail and skin care, footwear practices, and professional care seeking. Items are typically rated on a Likert scale, with higher scores indicating better self-care practices and greater confidence. The FCSOD has demonstrated strong reliability and validity, making it a valuable instrument for both clinical assessments and research studies aimed at improving foot health outcomes in older adults. Its user-friendly format also makes it suitable for elderly populations, whether self-administered or conducted via interviews.

SECONDARY OUTCOMES:
Foot Care Confidence Scale (FCCS) | through study completion, an average of 1 year
  The Foot Care Confidence Scale (FCCS) is a specialized instrument developed to measure an individual's self-efficacy, or confidence, in performing foot self-care activities to prevent diabetes-related foot complications. It assesses how confident patients feel about tasks such as inspecting their feet, maintaining proper hygiene, choosing appropriate footwear, and seeking professional help when necessary. The scale typically uses a Likert-type format, with higher scores indicating greater confidence in foot self-care abilities. The FCCS has demonstrated good reliability and validity in diabetic populations and is widely used in both clinical and research settings to guide interventions aimed at enhancing self-management and reducing the risk of serious foot problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: Yes